CLINICAL TRIAL: NCT05284955
Title: Efficacy of Pulmonary Pressure Guided Therapy in Stable Outpatients With Advanced Heart Failure - A Randomized Controlled Clinical Trial
Brief Title: Screening for Advanced Heart Failure IN Stable outPatientS - The SAINTS Study (SAINTS B)
Acronym: SAINTS B
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Collaborators: Novo Nordisk A/S (Industry); Abbott (Industry)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, Sponsor-Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH-SAINTS-B
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Advanced Heart Failure; Heart Failure With Reduced Ejection Fraction
Keywords: Advanced heart failure; Pulmonary pressure; Hemodynamics; Remote monitoring; Randomized controlled clinical trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CardioMEMS HF System group (Experimental): Pharmacological heart failure treatment guided by an implanted wireless pulmonary artery hemodynamic monitor (CardioMEMS HF system)
  Interventions: Device: CardioMEMS HF System
- Standard of care (Active Comparator): Standard heart failure medical treatment
  Interventions: Drug: Standard heart failure medical therapy

INTERVENTIONS:
Device: CardioMEMS HF System — The CardioMEMS HF System is a wireless pulmonary artery pressure monitor. We will use measurements from the device to guide medical heart failure therapy.
  Arms: CardioMEMS HF System group
Drug: Standard heart failure medical therapy — Standard heart failure medical therapy as recommended by guidelines.
  Arms: Standard of care

SUMMARY:
SAINTS B is a randomized, controlled, clinical trial. Patients identified with advanced heart failure in SAINTS A who are unwilling or unable to undergo heart transplantation or left ventricular assist device implantation will be invited to participate in this study. Included patients will be randomized in a 1:1 ratio to pharmacological HF treatment guided by an implanted wireless pulmonary artery hemodynamic monitor (CardioMEMS HF system) or usual care consisting of pharmacological HF treatment.

Patients randomized into the CardioMEMS arm will be implanted within 30 (Cardiomems group only) days from randomization. After randomization, patients in both the CardioMEMS and the control arm will be seen at the outpatient clinic at Rigshospitalet after one and 6 months. At the final clinical follow-up visit at 6 months, participants will perform a 6 minute walk test (6MWT), cardiopulmonary exercise test (CPET), fill out a quality of life questionnaire (Kansas City Cardiomyopathy Questionnaire (KCCQ)) and blood samples will be drawn. Patients in the CardioMEMS arm will be managed according to previously published protocols for pulmonary artery pressure optimization (generally mean pulmonary pressure 10-25 mmHg) (Ref 1).

DETAILED DESCRIPTION:
Data recording:

Data will be recorded in an online database using an electronic case report form. The investigators will use limits for accepted input, when applicable, on variables to minimize errors and specify which units the observations should be registered in. The investigators will perform quality controls two to four times per year of the database where new entries will be checked for accuracy and completeness.

Statistical considerations:

Sample size:

SAINTS A More than 3000 patients are followed in the HF clinics on Zealand including the greater Copenhagen region. The investigators plan to include 400 patients in the primary outcome analysis (SAINTS A) and hypothesize that 20% will fulfill the modified criteria for advanced HF.

SAINTS B Of the 80 patients identified in the main study, 60 can be expected to be available for randomization to CardioMEMS sensor implantation vs. clinical control. Mean (SD) KCCQ score in advanced HF is expected to be 64 with a standard deviation of 22, (Ref 2) and the investigators aim to see a 30% improvement with CardioMEMS. With a power of 80%, and an alpha of 5% this would require 21 patients in each group. With an expected dropout rate of 15%, a total sample of 48 patients would be required, and due to uncertainty of the estimate, the investigators aim to include 30 patients in each group. In a recent, large RCT on a HFrEF population without advanced HF, the baseline mean (SD) KCCQ score in the placebo group (n = 4112) were 68 (28,5) (Ref 3), which would require 30 patients in each arm for the same power calculation without correction for possible dropout.

Statistical analysis Descriptive statistics will be reported as mean +/- standard deviation (SD) or median (interquartile range (IQR)) depending on distribution. Comparisons between groups at baseline will be performed by unpaired t-tests for normally distributed continues variables, by the Mann-Whitney U test (Wilcoxon rank-sum) for non-normally distributed continuous variables and χ2 or Fisher's exact test for categorical variables.

The primary outcome of change in QoL assessed with the KCCQ from baseline to follow-up at 6 months between the intervention and control group will be tested with a paired t-test (and longitudinal data will be analyzed with linear mixed models with an indicator variable for the treatment group (Ref 4)). Secondary outcomes will be tested with paired and unpaired t-tests or Wilcoxon signed rank test depending on distribution, unadjusted χ2 test and a two-proportion z-test where appropriate. Treatment comparisons will be performed according to the intention to treat principle. Per protocol analyses will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Included in SAINTS A and fulfilling criteria for advanced HF (i.e., meeting primary endpoint for SAINTS A), although with a lower NT-proBNP cut-off level at ≥ 1000 pg/ml, but not referred for HTx or LVAD due to contraindications or patient preference
2. NYHA Functional class III
3. Be willing and able to upload pulmonary artery pressure information and comply with the follow-up requirements

Exclusion Criteria:

1. Systolic blood pressure < 90 mmHg
2. Chest circumference of > 165 cm if BMI is ≥35 kg/m2
3. Intolerance to all neurohormonal antagonists (i.e., intolerance to Angiotensin Converting Enzyme inhibitors (ACE-I), Angiotensin Receptor Blockers (ARBs), Angiotensin receptor II blocker - neprilysin inhibitor (ARNi), Mineralocorticoid Receptor Antagonists (MRA), hydralazine/isosorbide dinitrate, and betablockers)
4. Fluid overload with a maximum (or dose equivalent) diuretic intervention
5. Contraindications to 1-month dual antiplatelet therapy or anticoagulation therapy for post implantation
6. Significant congenital heart disease that has not been repaired and would prevent implantation of the CardioMEMS pulmonary artery sensor
7. Implanted with mechanical right heart valve(s)
8. Pregnant or planning to become pregnant in the next 12 months
9. An active, ongoing infection
10. History of current or recurrent (≥2 episodes within 5 years prior to consent) pulmonary emboli and/or deep vein thromboses

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life from baseline to 6 months follow-up measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ) score | 6 months from inclusion
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) score is a validated measure of quality of life in patients with HF. The range of the scale is 0-100, with higher values representing better quality of life.

SECONDARY OUTCOMES:
Mean pulmonary artery pressure and diastolic pulmonary artery pressure | 3 months from inclusion
  (only CardioMEMS arm)
Proportion reaching the preset pressure goal after 3 months | 3 months from inclusion
  (only Cardiomems arm)
Proportion reaching the preset pressure goal adjusted for baseline pulmonary artery pulsatility index | 3 months from inclusion
  (only Cardiomems arm)
Proportion of functioning devices | 6 months
  (only device arm)
Proportion of patients improving > 5 points on KCCQ score | 6 months
  Compared between intervention and control group
6 minute walk test distance in meters | 6 months
  Compared between intervention and control group
NTproBNP after 6 months | 6 months
  Compared between intervention and control group. N-terminal pro B-type natriuretic peptide (NTproBNP) in pg / ml
Estimated glomerular filtration rate (eGFR) in mL/min/1,73 m2 | 6 months
  Compared between intervention and control group
Time to hospitalization for heart failure | 6 months
Days spent alive out of hospital | 6 months
Mortality | 6 months
Number of out-patients visits | 6 months
Number of changes in loop diuretics and neurohomonal blockade | 6 months
Peak oxygen uptake in ml/kg/min | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, professor, PhD, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindenfeld J, Abraham WT, Maisel A, Zile M, Smart F, Costanzo MR, Mehra MR, Ducharme A, Sears SF, Desai AS, Paul S, Sood P, Johnson N, Ginn G, Adamson PB. Hemodynamic-GUIDEd management of Heart Failure (GUIDE-HF). Am Heart J. 2019 Aug;214:18-27. doi: 10.1016/j.ahj.2019.04.014. Epub 2019 May 3. No abstract available. PMID 31150790
- [Background] Aaronson KD, Stewart GC, Pagani FD, Stevenson LW, Palardy M, McNamara DM, Mancini DM, Grady K, Gorcsan J, Kormos R, Jeffries N, Taddei-Peters WC, Richards B, Khalatbari S, Spino C, Baldwin JT, Mann DL; REVIVAL Investigators. Registry Evaluation of Vital Information for VADs in Ambulatory Life (REVIVAL): Rationale, design, baseline characteristics, and inclusion criteria performance. J Heart Lung Transplant. 2020 Jan;39(1):7-15. doi: 10.1016/j.healun.2019.09.008. Epub 2019 Sep 14. PMID 31679943
- [Background] Teerlink JR, Diaz R, Felker GM, McMurray JJV, Metra M, Solomon SD, Adams KF, Anand I, Arias-Mendoza A, Biering-Sorensen T, Bohm M, Bonderman D, Cleland JGF, Corbalan R, Crespo-Leiro MG, Dahlstrom U, Echeverria LE, Fang JC, Filippatos G, Fonseca C, Goncalvesova E, Goudev AR, Howlett JG, Lanfear DE, Li J, Lund M, Macdonald P, Mareev V, Momomura SI, O'Meara E, Parkhomenko A, Ponikowski P, Ramires FJA, Serpytis P, Sliwa K, Spinar J, Suter TM, Tomcsanyi J, Vandekerckhove H, Vinereanu D, Voors AA, Yilmaz MB, Zannad F, Sharpsten L, Legg JC, Varin C, Honarpour N, Abbasi SA, Malik FI, Kurtz CE; GALACTIC-HF Investigators. Cardiac Myosin Activation with Omecamtiv Mecarbil in Systolic Heart Failure. N Engl J Med. 2021 Jan 14;384(2):105-116. doi: 10.1056/NEJMoa2025797. Epub 2020 Nov 13. PMID 33185990
- [Background] Rogers JG, Patel CB, Mentz RJ, Granger BB, Steinhauser KE, Fiuzat M, Adams PA, Speck A, Johnson KS, Krishnamoorthy A, Yang H, Anstrom KJ, Dodson GC, Taylor DH Jr, Kirchner JL, Mark DB, O'Connor CM, Tulsky JA. Palliative Care in Heart Failure: The PAL-HF Randomized, Controlled Clinical Trial. J Am Coll Cardiol. 2017 Jul 18;70(3):331-341. doi: 10.1016/j.jacc.2017.05.030. PMID 28705314